CLINICAL TRIAL: NCT01058408
Title: A Phase I Trial Using RAD001 With Weekly Cisplatin and Radiation Therapy in Patients With Locally Advanced Head and Neck Cancer
Brief Title: RAD001 With Weekly Cisplatin and Radiation Therapy in Patients With Locally Advanced Head and Neck Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Jochen Lorch, MD, Medical Oncology, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-342; CRAD001C4540T (Other: Novartis Pharmaceutical)
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Head and Neck Cancer
Keywords: advanced head and neck cancer; cisplatin; RAD001; radiation; HNSCC
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated; Everolimus; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rad001 with cisplatin (Experimental)
  Interventions: Radiation: Intensity modulated radiotherapy; Drug: RAD001; Drug: cisplatin

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy — Administered daily 5 days per week
  Other Names: IMRT
Drug: RAD001 — Taken orally once a day
Drug: cisplatin — Administered intravenously once a week

SUMMARY:
RAD001 is approved by the U.S Food and Drug Administration (FDA) to treat advanced kidney cancer. This drug has also been used in other research studies to evaluate its effectiveness in other cancers. Information from these research studies suggests that RAD001 may help to decrease the growth and development of tumor cells by reducing the blood supply that tumors need to grow. In this research study, we are trying to determine the safety of RAD001 when given to people with locally advanced head and neck cancer in combination with cisplatin and radiation. We are also looking for the highest dose of RAD001 that can be given to people safely.

DETAILED DESCRIPTION:
* Most patients receiving treatment for head and neck cancer will develop difficulty swallowing food and drinking liquids during the course of therapy. For this reason, it will be recommended that a PEG (percutaneous endoscopic gastrostomy) tube be placed in the participants stomach prior to undergoing the study regimen. This is to help maintain weight and nutritional health.
* Since we are looking for highest dose of the study drug that can be administered safely without severe or unmanageable side effects, not everyone who participates will receive the same dose of RAD001 or cisplatin.
* The study regimen will last for seven weeks. During each week of study participation the following will occur: Radiation will be administered each weekday (5 days per week). Cisplatin will be given intravenously at the start of each week. RAD001 will be given to the participant to take at home. Participants will take the study drug once a day in the morning starting on day 1.
* A history and physical exam will be performed weekly while participant's are receiving radiation treatment. Blood tests for routine laboratory testing will be performed weekly.
* Each month for the first two months after participants finish radiation therapy and stop taking RAD001 and cisplatin, they will have a physical ezam, a neurologic exam, and blood tests. X-rays, a CT, MRI and/or PET scans will also be performed a the two month visit. After the first two months, follow-up will continue every 1-2 months for the first year. Additionally, every 6 months for the first two years, follow-up visits will include an assessment of speech and swallowing functions along with X-rays, CT, MRI and/or PET scans.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage III/IV, locally advanced, biopsy proven squamous cell cancer of the head and neck who are planned to undergo chemoradiation as their primary treatment with curative intent. Patients with oropharynx, hypopharynx, larynx primaries, nasopharynx as well as those with documented SCC of the cervical lymph nodes, with unknown primaries, are eligible.
* Patients must have at least evaluable disease and one measurable site of disease according to RECIST criteria is desirable.
* 18 years of age or older
* Minimum of two weeks since any major surgery
* WHO performance status of 2 or less
* Adequate bone marrow, liver, and renal function as outlined in the protocol

Exclusion Criteria:

* Presence of distant metastatic disease
* Prior chemotherapy
* Prior radiation to the head and neck or adjacent anatomical site
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Other malignancies within the past 3 years except for adequately treated carcinoma of the thyroid, cervix or basal or squamous cell carcinomas of the skin
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Uncontrolled diabetes mellitus
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001
* Patients with an active, bleeding diathesis or on oral anti-vitamin K medication
* Women who are pregnant or breastfeeding, or women/men able to conceive and unwilling to practice an effective method of birth control
* Patients who have received prior treatment with an mTOR inhibitor
* Patients with a known hypersensitivity to RAD001 or other rapamycins or to its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the maximum tolerated dose (MTD) and safety of the RAD001 in combination with weekly cisplatin and radiation in patients with locally advanced HNSCC. | 2 years

SECONDARY OUTCOMES:
Obtain preliminary results on efficacy of the RAD001, cisplatin and radiation therapy combination in patients with locally advanced HNSCC. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Lorch, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States